CLINICAL TRIAL: NCT02586155
Title: A Phase III Multi-Center, Double-Blind, Randomized, Parallel Group, Placebo-Controlled Clinical Trial in High-Risk Type 2 Diabetes Mellitus (T2DM) Subjects With Coronary Artery Disease (CAD) to Determine Whether Bromodomain Extraterminal Domain (BET) Inhibition Treatment With RVX000222 Increases the Time to Major Adverse Cardiovascular Events (MACE)
Brief Title: Effect of RVX000222 on Time to Major Adverse Cardiovascular Events in High-Risk T2DM Subjects With CAD
Acronym: BETonMACE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Resverlogix Corp (Industry)
Collaborators: PPD Development, LP (Industry); ICON plc (Industry); Medidata Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RVX222-CS-015
Record Dates: First submitted 2015-10-21; First posted 2015-10-26 (Estimated); Results first posted 2021-08-20 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-07

CONDITIONS: Diabetes Mellitus, Type 2; Coronary Artery Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Coronary Artery Disease | interventions — apabetalone; Atorvastatin; Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- High-Intensity statin therapy+RVX000222 (Experimental): Daily dose 100 mg capsule b.i.d. with high-intensity statin therapy (atorvastatin or rosuvastatin)
  Interventions: Drug: Apabetalone; Drug: Atorvastatin; Drug: Rosuvastatin
- High-Intensity statin therapy+Placebo (Active Comparator): Placebo (for RVX000222 100 mg capsule) b.i.d. with high-intensity statin therapy (atorvastatin or rosuvastatin)
  Interventions: Drug: Placebo; Drug: Atorvastatin; Drug: Rosuvastatin

INTERVENTIONS:
Drug: Apabetalone — 100 mg capsule
  Other Names: RVX000222
  Arms: High-Intensity statin therapy+RVX000222
Drug: Placebo — Capsule manufactured to mimic RVX000222 100 mg capsule
  Other Names: Placebo (for RVX000222)
  Arms: High-Intensity statin therapy+Placebo
Drug: Atorvastatin — High-Intensity Statin
  Other Names: Lipitor
Drug: Rosuvastatin — High-Intensity Statin
  Other Names: Crestor

SUMMARY:
The purpose of this study is to determine whether bromodomain extraterminal domain (BET) inhibition treatment with RVX000222 in high-risk type 2 diabetes mellitus patients with coronary artery disease increases the time to major adverse cardiovascular events.

DETAILED DESCRIPTION:
The majority (75%) of deaths in subjects with diabetes mellitus (DM) are due to atherosclerotic cardiovascular disease (CVD). Recent studies suggest a major adverse cardiovascular event (MACE) rate of >11% over 18 months in type 2 diabetes mellitus (T2DM) despite a baseline LDL-C of <2.1 mmol/L. Bromodomains (BRDs) are a family of evolutionary conserved protein-interaction modules that play key functions in chromatin organization and regulation of gene transcription. One recognized family of bromodomain-containing proteins is the bromodomain and extra-terminal (BET) family. BET inhibition represents a novel, epigenetic approach to treat CAD.

RVX000222 affects biological processes important in atherosclerosis and acute coronary events via selective inhibition of BET proteins. RVX000222 is available as a capsule formulation with standard excipients and established stability.

The BETonMACE study will focus on prevention of subsequent MACE in subjects with CAD and DM with high intensity statin therapy as co-medication.

ELIGIBILITY:
Inclusion Criteria:

• ACS event of either unstable angina or myocardial infarction 7-90 days prior Visit 1:

Unstable angina: for a qualifying unstable angina event, each of components (a), (b), and (c) must be satisfied: a.) Characteristic ischemic pain or discomfort in chest/associated referral areas, occurring at rest/with minimal exertion b.) ECG changes consistent with acute myocardial ischemia based on new/presumed ST elevation/depression or T-wave inversion c.) Objective evidence of obstructive CAD based on 1+ of the following: i. New/presumed new evidence of myocardial ischemia/infarction by perfusion imaging ii. New/presumed new regional wall motion abnormality iii. Current evidence of at least 1 epicardial coronary artery stenosis ≥70% by coronary angiography iv. Need for coronary revascularization for the index ACS event, including a percutaneous coronary intervention (PCI) with or without coronary stenting.

Prior MI 7-90 days prior screening treated with or without a percutaneous coronary intervention (PCI). For a qualifying event of MI 2 of the following 3 criteria must be satisfied: a.) Characteristic ischemic chest pain/pain in associated referral areas b.) Dynamic elevation of troponin T/I or CKMB if troponinT/I is unavailable at local lab (at least >ULN for lab) c.) Development of new Q-waves in ≥2 adjacent ECG leads or development of new dominant R wave in V1

* Documented diagnosis of T2DM (1+ of the following criteria): Documented history of T2DM, History of taking diabetes medication, and/or HbA1c ≥6.5% at Visit 1
* For males HDL-C<40 mg/dL(1.04 mmol/L), for females HDL-C<45 mg/dL(1.17 mmol/L) at Visit 1
* Subjects currently not on high intensity statin therapy could start rosuvastatin at Visit 1 and those currently on therapy besides atorvastatin/rosuvastatin can be switched to rosuvastatin at Visit 1
* Female subjects of non-childbearing potential (post-surgical sterilization/post-menopausal) or if childbearing potential have neg urine pregnancy test and be willing and able to use non-hormonal birth control (non-hormonal IUD, condom or diaphragm) or remain abstinent from Screening to Follow-up Visit
* Give signed informed consent

Exclusion Criteria:

* Heart disease which will w/in 90 days of Visit 1 likely need coronary bypass, PCI, cardiac transplantation, surgical repair and/or replacement
* Previous/current diagnosis of severe heart failure or documented LVEF<25% determined by contrast left ventriculography, radionuclide ventriculography or echocardiography. Absence of LVEF measurement in subject w/out a previous/current diagnosis of heart failure does not exclude entry into study
* Evidence of cardiac EP instability incl. history of uncontrolled ventricular arrhythmias, atrial fibrillation/flutter or supraventricular tachycardias w/ a ventricular response HR>100bpm at rest w/in 4 wks prior Visit 1
* CABG w/in 90 days prior Visit 1
* Evidence of severe renal impairment as determined by either eGFR<30 mL/min/1.7m2 at Visit 1 or current need for dialysis
* Uncontrolled hypertension defined as 2 consecutive measurements of sitting BP of systolic>180 mmHg or diastolic>100 mmHg at Visit 1
* Treatment w/ immunosuppressants w/in 12 mos prior Visit 1
* Use of fibrates at any dose or niacin/nicotinic acid 250+ mg w/in 30 days prior Visit 1
* Known allergy/sensitivity to any ingredient in IMP
* History of intolerance to atorvastatin/rosuvastatin
* Triglycerides>400 mg/dL (4.52 mmol/L) at Visit 1
* Any medical/surgical condition which might significantly alter absorption, distribution, metabolism or excretion of medication
* Evidence of cirrhosis from liver imaging/biopsy, history of hepatic encephalopathy, esophageal/gastric varices, active hepatitis or prior porta-caval shunt procedure or a Child-Pugh score of ≥5 points
* ALT/AST>1.5xULN by central lab at Visit 1
* Tot. bilirubin>ULN by central lab at Visit 1
* History of malignancy of any organ syst treated/untreated w/in the past 2 yrs whether or not there is evidence of local recurrence/metastases except localized basal skin cell carcinoma
* History/evidence of drug/alcohol abuse w/in 12 mos of Visit 1
* Pregnancy
* Any condition which may place subject at higher risk from his/her participation in the study or is likely to prevent subject from completing/complying w/ requirements of study
* Use of other investigational drugs and devices w/in 30 days or 5 half-lives of Visit 1, whichever is longer
* History of noncompliance to medical regimens or unwillingness to comply w/ study protocol
* Any condition that would confound the evaluation/interpretation of efficacy and/or safety data
* Persons directly involved in execution of this protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2425 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kausik Ray, MD, Study Chair — Imperial College London
Locations (214):
- Argentina (36):
  - Instituto de Investigaciones Clinicas Bahia Blanca, Bahía Blanca
  - Bioclinica Buenos Aires, Buenos Aires
  - Centro Privado de Enfermedades Cardiovasculares, Buenos Aires
  - Consultorios Asociados Endocronología E Investigación Clínica Aplicada, Buenos Aires
  - Instituto Cardiovascular de Buenos Aires, Buenos Aires
  - Sanatorio Guemes, Buenos Aires
  - Clinica Coronel Suarez, Coronel Suárez
  - Instituto de Cardiologia de Corrientes Juana Francisca Cabral, Corrientes
  - CEMAIC, Córdoba
  - Centro Médico Colón, Córdoba
  - Centro Médico Luquez, Córdoba
  - Clínica Privada Del Prado Sociedad de Responsabilidad Limitada, Córdoba
  - Fundación Clínica Colombo, Córdoba
  - Hospital Cordoba, Córdoba
  - Hospital San Roque, Córdoba
  - Instituto Del Corazón, Córdoba
  - Instituto Modelo de Cardiologia, Córdoba
  - Instituto Médico DAMIC, Córdoba
  - Ipac Caraffa, Córdoba
  - Sanatorio Allende, Córdoba
  - Centro Médico Libertad, Haedo
  - CIMEL, Lanús
  - Instituto de Investigaciones Clínicas Mar Del Plata, Mar del Plata
  - Hospital Central, Mendoza
  - DIM Clinica Privada, Ramos Mejía
  - Instituto de Hematologia Y Medicina Clinica, Rosario
  - Sanatorio Britanico de Rosario, Rosario
  - Prevencion Cardio Vascular, Salta
  - Grupo Medico Alem, San Isidro
  - Bioclinica Tucumán, San Miguel de Tucumán
  - Centro Modelo de Cardiologia, San Miguel de Tucumán
  - Investigaciones Clinicas Tucuman, San Miguel de Tucumán
  - Centro de Investigaciones Clínicas Del Litoral SRL, Santa Fe
  - Sanatorio San Francisco, Santiago del Estero
  - Clínica FUSAVIM Privada, Villa María
  - Instituto de Investigaciones Clínicas Zárate, Zárate
- Flinders Medical Centre, Bedford Park, Australia
- Belgium (3):
  - ZNA Middelheim, Antwerp
  - Imelda VZW, Bonheiden
  - AZ Turnhout, Turnhout
- Bulgaria (14):
  - Multiprofile Hospital For Active Treatment Dr Tota Venkova, Gabrovo
  - Multiprofile Hospital for Active Treatment - Prof. Dr. Paraskev Stoyanov AD, Lovech
  - Multiprofile Hospital For Active Treatment - Pazardzhik AD, Pazardzhik
  - University Multiprofile Hospital for Active Treatment - Dr. Georgi Stranski EAD, Pleven
  - Multiprofile Hospital For Active Treatment - Dr. Bratan Shukerov AD, Smolyan
  - Acibadem City Clinic Multiprofile Hospital for Active Treatment Tokuda, Sofia
  - City Clinic University Multiprofile Hospital for Active Treatment EOOD, Sofia
  - Medical Center Kardiohelp EOOD, Sofia
  - Second Multiprofile Hospital for Active Treatment Sofia, Sofia
  - Synexus Affiliate - Diagnostic and Consulting Center Ascendent, Sofia
  - University Multiprofile Hospital for Active Treatment Aleksandrovska EAD, Sofia
  - University Multiprofile Hospital for Active Treatment and Emergency Medicine N. I. Pirogov EAD, Sofia
  - Medical Center Orfey OOD, Stara Zagora
  - Multiprofile Hospital for Active Treatment Sveta Marina EAD, Varna
- Croatia (6):
  - General Hospital Karlovac, Karlovac
  - Special Hospital for medicinal rehabilitation Krapinske Toplice, Krapinske Toplice
  - Clinical Hospital Osijek, Osijek
  - General Hospital Dr Josip Bencevic, Slavonski Brod
  - General Hospital Virovitica, Virovitica
  - Clinical Hospital Sveti duh, Zagreb
- Germany (9):
  - DRK Kliniken Berlin Westend, Berlin
  - Medizinisches Versorgungszentrum am Küchwald GmbH, Chemnitz
  - Zentrum für Klinische Prüfung in der Facharztzentrum Dresden Neustadt Gbr, Dresden
  - Katholisches Krankenhaus St. Johann Nepomuk, Erfurt
  - Heidelberger Praxisklinik für Kardiologie, Heidelberg
  - Klinikum Hoyerswerda, Hoyerswerda
  - Studienzentrum Dr.Appel, Kassel
  - Asklepios Klinik Langen, Langen
  - Klinikum Leverkusen GmbH, Leverkusen
- Hungary (17):
  - Bajai Szent Rókus Kórház, Baja
  - Grof Tisza Istvan Korhaz Berettyoujfalu, Berettyóújfalu
  - Bajcsy-Zsilinszky Korhaz es Rendelointezet, Budapest
  - Del-pesti Centrumkorhaz- Orszagos Hematologiai és Infektologiai Intezet, Budapest
  - Gottsegen Gyorgy Orszagos Kardiologiai Intezet, Budapest
  - Magyar Honvédség Egészségügyi Központ, Budapest
  - Semmelweis Egyetem, Budapest
  - Synexus (DRS) - Synexus Magyarország Kft. Budapest, Budapest
  - Szent Margit Korhaz, Budapest
  - Szent Rókus Kórház és Intézményei, Budapest
  - Selye János Kórház, Komárom
  - TaNaMed Kft., Mosonmagyaróvár
  - Kanizsai Dorottya Kórház, Nagykanizsa
  - Coromed-SMO Kft., Pécs
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont, Szeged
  - Tolna Megyei Balassa János Kórház, Szekszárd
  - Fejer Megyei Szent Gyorgy Egyetemi Oktato Korhaz, Székesfehérvár
- Israel (20):
  - Barzilai Medical Center, Ashkelon
  - Soroka University Medical Centre, Beersheba
  - Hillel Yaffe Medical Center, Hadera
  - Bnei Zion Medical Center, Haifa
  - Lady Davis Carmel Medical Center, Haifa
  - Linn Medical Center Clalit Health Services, Haifa
  - Rambam Medical Center, Haifa
  - Edith Wolfson Medical Center, Holon
  - Hadassah University Hospital Ein Kerem, Jerusalem
  - Hadassah University Hospital Mount Scopus, Jerusalem
  - Shaare Zedek Medical Center, Jerusalem
  - Meir Medical Center, Kefar Sava
  - Galilee Medical Center, Nahariya
  - Nazareth EMMS Hospital, Nazareth
  - Chaim Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - ZIV Medical Center, Safed
  - Clalit Health Medical Center, Tel Aviv
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Baruch Padeh Poriya Medical Center, Tiberias
- Mexico (25):
  - Fundacion Cardiovascular de Aguascalientes AC, Aguascalientes
  - Hospital Cardiológica Aguascalientes, Aguascalientes
  - Investigacion en Salud y Metabolismo S.C., Chihuahua City
  - Centro Para el Desarrollo de la Medicina y de Asistencia Especializada SC, Culiacán
  - Centro de Investigacion y Atencion de Diabetes, Endocrinologia y Nutricion, Durango
  - Arechavaleta Granell Maria del Rosario, Guadalajara
  - Centro de Investigacion Medica Biologica Y de Terapia Avanzada SC, Guadalajara
  - Unidad de Investigacion Clinica Cardiometabolica de Occidente SC, Guadalajara
  - Hospital Angeles Leon, León
  - Centro de Investigación Biomedica y Farmaceutica, Mexico City
  - Clinica Integral del Paciente Diabetico y Obeso, Mexico City
  - Fundación de Atención e Investigación Médica Lindavista S.C., Mexico City
  - Sanatorio y Servicios Médicos Obregón S.A. de C.V., Mexico City
  - Centro de Desarrollo Biomédico, Mérida
  - Instituto Cardiovascular de Monclova, Monclova
  - Hospital Universitario Dr. Jose Eleuterio González, Monterrey
  - IMED Internal Medicine Clin Trials, Monterrey
  - Unidad de Investigación Clínica En Medicina SC, Monterrey
  - Diabetes Total, S.A de C.V., Pachuca
  - Investigacion Biomedica Aplicada de Hidalgo S.A. de C.V., Pachuca
  - Cardioarritmias e Investigación S.C., San Luis Potosí City
  - Hospital Central Dr Ignacio Morones Prieto, San Luis Potosí City
  - INBIOMEDYC Toluca, Toluca
  - Centro de Alta Especialidad Dr. Rafael Lucio, Veracruz
  - Dr. Humberto Alvarez Lopez, Zapopan
- Netherlands (3):
  - Meander Medisch Centrum, Amersfoort
  - OLVG locatie Oost, Amsterdam
  - VU Medisch Centrum, Amsterdam
- Poland (21):
  - Podlaski Osrodek Kardiologii Poradnia Prywatna, Bialystok
  - Malopolskie Centrum Sercowo-Naczyniowe, Chrzanów
  - Polsko-Amerykanskie Kliniki Serca, Dąbrowa Górnicza
  - Gabinet Kardiologiczno-Internistyczny, Gdynia
  - Niepubliczny Zaklad Opieki Zdrowotnej Centrum Uslug Medycznych Promont-Med., Kielce
  - Diamond Clinic, Krakow
  - Szpital Specjalistyczny im. Jozefa Dietla w Krakowie, Krakow
  - Zespol Przychodni Specjalistycznych DIAB-END-COR Sp. z o.o., Krakow
  - Prywatna Praktyka Lekarska MAZ-MEDICA Maciej R.Mazurkiewicz, Lodz
  - Uniwersytecki Szpital Kliniczny im. Wojskowej Akademii Medycznej Centralny Szpital Weteranow, Lódz
  - Polsko-Amerykanskie Kliniki Serca, Nysa
  - Pro Corde, Dom Medyczny, Opole
  - Medicome Sp. z o.o., Oświęcim
  - Rodzinne Centrum Zdrowia, Otwock
  - Niepubliczny Zaklad Opieki Zdrowotnej Specjalistyczna Przychodnia Lekarska "MEDIKARD", Płock
  - Niepubliczny Zaklad Opieki Zdrowotnej Centrum Medyczne SBB, Tarnobrzeg
  - Centrum Medyczne doktorA, Warsaw
  - Instytut Kardiologii im Prymasa Tysiaclecia Kardynala Stefana Wyszynskiego, Warsaw
  - Niepubliczny Zaklad Opieki Zdrowotnej AURUM, Warsaw
  - Centrum Kardiologiczne Pro Corde Sp. z o.o. Niepubliczny Zaklad Opieki Zdrowotnej, Wroclaw
  - Wro Medica, Wroclaw
- Russia (19):
  - City Clinical Hospital #6, Chelyabinsk
  - Federal Budget Healthcare Institution Medici - sanitary unit of Ministry of internal affairs of Russ, Kemerovo
  - Research Institute of Complex Cardiovascular Pathology, Kemerovo
  - Krasnodar Regional Clinical Hospital #2, Krasnodar
  - Moscow City State Budgetary Healthcare Institution City Clinical Hospital named after V.V. Veresayev, Moscow
  - Russian Cardiology Research and Production Center, Moscow
  - City Hospital 13, Nizhny Novgorod
  - State Budgetary Healthcare Institution of Novosibirsk Region City Clinical Hospital No. 19, Novosibirsk
  - Republican Hospital n.a. V.A. Baranov, Petrozavodsk
  - Municipal Budgetary Healthcare Institution City Emergency Hospital, Rostov-on-Don
  - International Medical Center SOGAZ, Saint Petersburg
  - North-West State Medical University n.a. I.I. Mechnikov, Saint Petersburg
  - St Petersburg City Outpatient Clinic #109, Saint Petersburg
  - Saratov State Medical University, Saratov
  - State Healthcare Institution Regional Clinical Cardiologic Dispensary, Saratov
  - City Hospital #4, Sochi
  - Research Cardiology Institute of Tomsk Scientific Center of RAMS Siberian Branch, Tomsk
  - State Budgetary Healthcare Institution of Vladimir Region City Hospital No. 4, Vladimir
  - Ural State Medical University, Yekaterinburg
- Serbia (15):
  - Clinical Center of Serbia, Belgrade
  - Clinical Hospital Centar Zvezdara, Belgrade
  - Clinical Hospital Center Bezanijska Kosa, Belgrade
  - Clinical Hospital Centre Zemun, Belgrade
  - Euromedik, Belgrade
  - Institute of Cardiovascular Diseases Dedinje, Belgrade
  - KBC Dr Dragisa Misovic Dedinje, Belgrade
  - Military Medical Academy, Belgrade
  - Institute of Cardiovascular Diseases of Vojvodina, Kamenitz
  - Clinical Center Kragujevac, Kragujevac
  - Clinical Center Nis, Niš
  - Institute Niska Banja, Niška Banja
  - Clinical Centre of Vojvodina, Novi Sad
  - General Hospital Uzice, Užice
  - Health Center Zajecar, Zaječar
- Slovakia (12):
  - ALIAN, s.r.o, Bardejov
  - CARDIOCONSULT, s.r.o., Bratislava
  - Univerzitna nemocnica Bratislava, Bratislava
  - Kardio-Onkologia, s.r.o., Dolný Kubín
  - CARDIO D&R, s.r.o. Kosice, Košice
  - Zeleznicne zdravotnictvo Kosice, s.r.o., Košice
  - KARDIOMED s.r.o., Lučenec
  - MEDI M&M s.r.o., Moldava nad Bodvou
  - Nemocnica s poliklinikou Nove Mesto nad Vahom n.o., Nové Mesto nad Váhom
  - Cardioinvest s. r. o., Nové Zámky
  - DIAB s.r.o., Rožňava
  - MEDIVASA, s.r.o., Žilina
- Taiwan (13):
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Mackay Memorial Hospital-Taipei branch, New Taipei City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Cathay General Hospital, Taipei
  - Chi Mei Medical Center, Taipei
  - Far Eastern Memorial Hospital, Taipei
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Medical Foundation Linkou Branch (Clinical Research Center), Taoyuan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ray KK, Nicholls SJ, Buhr KA, Ginsberg HN, Johansson JO, Kalantar-Zadeh K, Kulikowski E, Toth PP, Wong N, Sweeney M, Schwartz GG; BETonMACE Investigators and Committees. Effect of Apabetalone Added to Standard Therapy on Major Adverse Cardiovascular Events in Patients With Recent Acute Coronary Syndrome and Type 2 Diabetes: A Randomized Clinical Trial. JAMA. 2020 Apr 28;323(16):1565-1573. doi: 10.1001/jama.2020.3308. PMID 32219359
- [Derived] Schwartz GG, Nicholls SJ, Toth PP, Sweeney M, Halliday C, Johansson JO, Wong NCW, Kulikowski E, Kalantar-Zadeh K, Ginsberg HN, Ray KK. Relation of insulin treatment for type 2 diabetes to the risk of major adverse cardiovascular events after acute coronary syndrome: an analysis of the BETonMACE randomized clinical trial. Cardiovasc Diabetol. 2021 Jun 22;20(1):125. doi: 10.1186/s12933-021-01311-9. PMID 34158057
- [Derived] Haarhaus M, Gilham D, Kulikowski E, Magnusson P, Kalantar-Zadeh K. Pharmacologic epigenetic modulators of alkaline phosphatase in chronic kidney disease. Curr Opin Nephrol Hypertens. 2020 Jan;29(1):4-15. doi: 10.1097/MNH.0000000000000570. PMID 31725015
- [Derived] Ray KK, Nicholls SJ, Ginsberg HD, Johansson JO, Kalantar-Zadeh K, Kulikowski E, Toth PP, Wong N, Cummings JL, Sweeney M, Schwartz GG. Effect of selective BET protein inhibitor apabetalone on cardiovascular outcomes in patients with acute coronary syndrome and diabetes: Rationale, design, and baseline characteristics of the BETonMACE trial. Am Heart J. 2019 Nov;217:72-83. doi: 10.1016/j.ahj.2019.08.001. Epub 2019 Aug 9. PMID 31520897
- [Derived] Gilham D, Tsujikawa LM, Sarsons CD, Halliday C, Wasiak S, Stotz SC, Jahagirdar R, Sweeney M, Johansson JO, Wong NCW, Kalantar-Zadeh K, Kulikowski E. Apabetalone downregulates factors and pathways associated with vascular calcification. Atherosclerosis. 2019 Jan;280:75-84. doi: 10.1016/j.atherosclerosis.2018.11.002. Epub 2018 Nov 14. PMID 30476723

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High-Intensity Statin Therapy+RVX000222 | High-Intensity Statin Therapy+Placebo
Started | 1215 | 1210
Final Number Randomized | 1212 | 1206
Completed | 1088 | 1083
Not Completed | 127 | 127
Not completed — Adverse Event | 2 | 3
Not completed — Withdrawal by Subject | 31 | 24
Not completed — Lost to Follow-up | 7 | 13
Not completed — Death | 61 | 72
Not completed — Other reasons | 26 | 15

BASELINE CHARACTERISTICS:
Population: Of the initial 1215 participants randomized into the High-Intensity statin therapy+RVX000222 group, 3 were randomized in error. Of the initial 1210 participants randomized into the High-Intensity statin therapy+placebo group, 4 were randomized in error.
Groups:
- Total: Total of all reporting groups
Arm/Group | High-Intensity Statin Therapy+RVX000222 | High-Intensity Statin Therapy+Placebo | Total
Number analyzed (Participants) | 1212 | 1206 | 2418
Age, Continuous [Median (Full Range); unit: years] | 62.0 [33.0 to 85.0] | 62.0 [31.0 to 88.0] | 62.0 [31.0 to 88.0]
Age, Customized [Count of Participants; unit: Participants]
  ≤65 years | 816 | 772 | 1588
  >65 years | 396 | 434 | 830
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 305 | 313 | 618
  Male | 907 | 893 | 1800
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 27 | 31 | 58
  Asian | 20 | 19 | 39
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1063 | 1056 | 2119
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 102 | 100 | 202
Body weight [Median (Full Range); unit: kilograms (kg)] — Population: Body weight data is missing for some subjects
  kilograms (kg)
    number analyzed (Participants) | 1210 | 1206 | 2416
    (all) | 85.75 [47.5 to 162.0] | 85.90 [43.6 to 160.0] | 85.90 [43.6 to 162.0]
Body-mass index (BMI) [Median (Full Range); unit: kg/m2] — Population: Body-mass index (BMI) data missing for some subjects
  kg/m2
    number analyzed (Participants) | 1208 | 1206 | 2414
    (all) | 29.589 [20.04 to 53.46] | 29.585 [18.33 to 51.17] | 29.585 [18.33 to 53.46]

OUTCOME MEASURES:

1. Primary Outcome: Incidence of First Occurrence of Adjudication-confirmed Narrowly Defined MACE
Description: Incidence of first occurrence of MACE narrowly defined as a single composite endpoint of Cardiovascular (CV) Death (including undetermined cause of death) or Non-fatal Myocardial Infarction (MI) or Stroke. If a subject has multiple events, only the first event contributing to the composite endpoint is counted.
Time Frame: 120 weeks
Measure: Number; unit: events
Arm/Group | High-Intensity Statin Therapy+RVX000222 | High-Intensity Statin Therapy+Placebo
Number analyzed (Participants) | 1212 | 1206
events
  CV Death | 34 | 42
  Non-fatal MI | 76 | 92
  Stroke | 15 | 15
Statistical Analysis 1: Comparison: High-Intensity Statin Therapy+RVX000222 vs High-Intensity Statin Therapy+Placebo; Test type: Superiority; p = 0.1070, Stratified long-rank; Cox Proportional Hazard = 0.823, 95% CI 2-sided [0.649 to 1.044]

2. Secondary Outcome: Incidence of First Occurrence of Adjudication-confirmed Broadly Defined MACE
Description: First occurrence of MACE broadly defined as a single composite endpoint of Cardiovascular Death (CVD) (including undetermined cause of death) or Non-fatal Myocardial Infarction (MI), Stroke, or Hospitalization for CVD events (including unstable angina and evidence of new or presumed new progressive obstructive coronary disease or emergency revascularization procedures at any time and urgent revascularization procedures ≥30 days after the index event as defined by Hicks et al., 2014) . If a subject has multiple events, only the first event contributing to the composite endpoint is counted.
Time Frame: 120 weeks
Measure: Number; unit: events
Arm/Group | High-Intensity Statin Therapy+RVX000222 | High-Intensity Statin Therapy+Placebo
Number analyzed (Participants) | 1212 | 1206
events
  CV Death | 33 | 42
  Non-fatal MI | 74 | 91
  Hospitalization for CVD events | 22 | 18
  Stroke | 15 | 15
Statistical Analysis 1: Comparison: High-Intensity Statin Therapy+RVX000222 vs High-Intensity Statin Therapy+Placebo; Test type: Superiority; p = 0.1495, Stratified long-rank; Cox Proportional Hazard = 0.849, 95% CI 2-sided [0.679 to 1.061]

3. Secondary Outcome: Incidence of Hospitalization for Congestive Heart Failure (CHF)
Time Frame: 120 weeks
Measure: Number; unit: events
Arm/Group | High-Intensity Statin Therapy+RVX000222 | High-Intensity Statin Therapy+Placebo
Number analyzed (Participants) | 1212 | 1206
events | 29 | 48
Statistical Analysis 1: Comparison: High-Intensity Statin Therapy+RVX000222 vs High-Intensity Statin Therapy+Placebo; Test type: Superiority; p = 0.03, Stratified long-rank; Hazard Ratio (HR) = 0.59, 95% CI 2-sided [0.38 to 0.94]

4. Secondary Outcome: Incidence of All-cause Mortality
Time Frame: 120 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | High-Intensity Statin Therapy+RVX000222 | High-Intensity Statin Therapy+Placebo
Number analyzed (Participants) | 1212 | 1207
Participants | 61 | 72
Statistical Analysis 1: Comparison: High-Intensity Statin Therapy+RVX000222 vs High-Intensity Statin Therapy+Placebo; Test type: Superiority; p = 0.44, Stratified long-rank; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.62 to 1.24]

5. Secondary Outcome: Change in Apolipoprotein A1 (ApoA-I) Concentration From Baseline Over Time Within and Between Treatment Groups
Time Frame: 120 weeks
Population: A select subset of subjects were analyzed for ApoA-I, Subject data is missing across time points.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | High-Intensity Statin Therapy+RVX000222 | High-Intensity Statin Therapy+Placebo
Number analyzed (Participants) | 243 | 238
mg/dL
  Baseline | 119.0 [110.0 to 130.0] | 117.5 [108.0 to 128.0]
  Visit 11 (Week 24): number analyzed (Participants) | 216 | 203
  Visit 11 (Week 24) | 128.0 [118.5 to 138.5] | 125.0 [114.0 to 138.0]
  Visit 14 (Week 52): number analyzed (Participants) | 207 | 201
  Visit 14 (Week 52) | 129.0 [118.0 to 141.0] | 124.0 [114.0 to 136.0]
  Visit 16 (Week 76): number analyzed (Participants) | 162 | 166
  Visit 16 (Week 76) | 132.0 [119.0 to 146.0] | 125.0 [112.0 to 136.0]
  Visit 18 (Week 100): number analyzed (Participants) | 112 | 117
  Visit 18 (Week 100) | 131.0 [119.0 to 142.5] | 125.0 [115.0 to 138.0]
  Last Visit on Treatment (LVT): number analyzed (Participants) | 174 | 184
  Last Visit on Treatment (LVT) | 132.5 [120.0 to 147.0] | 129.0 [115.5 to 141.0]
  Follow-up: number analyzed (Participants) | 165 | 171
  Follow-up | 131.0 [119.0 to 146.0] | 127.0 [116.0 to 143.0]

6. Secondary Outcome: Change in Apolipoprotein B (apoB) Concentration From Baseline Over Time Within and Between Treatment Groups
Time Frame: 120 weeks
Population: A select subset of subjects were analyzed for ApoB, Subject data is missing across time points.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | High-Intensity Statin Therapy+RVX000222 | High-Intensity Statin Therapy+Placebo
Number analyzed (Participants) | 243 | 238
mg/dL
  Baseline | 66.0 [54.0 to 80.0] | 66.0 [53.0 to 80.0]
  Visit 11 (Week 24): number analyzed (Participants) | 216 | 203
  Visit 11 (Week 24) | 68.5 [55.0 to 80.5] | 68.0 [53.0 to 86.0]
  Visit 14 (Week 52): number analyzed (Participants) | 207 | 201
  Visit 14 (Week 52) | 70.0 [59.0 to 84.0] | 68.0 [56.0 to 85.0]
  Visit 16 (Week 76): number analyzed (Participants) | 162 | 166
  Visit 16 (Week 76) | 70.5 [58.0 to 87.0] | 69.0 [55.0 to 89.0]
  Visit 18 (Week 100): number analyzed (Participants) | 112 | 117
  Visit 18 (Week 100) | 70.5 [59.0 to 85.0] | 72.0 [58.0 to 89.0]
  Last Visit on Treatment (LVT): number analyzed (Participants) | 174 | 184
  Last Visit on Treatment (LVT) | 68.0 [56.0 to 85.0] | 72.0 [57.5 to 89.0]
  Follow-up: number analyzed (Participants) | 165 | 171
  Follow-up | 70.0 [57.0 to 86.0] | 71.0 [57.0 to 89.0]

7. Secondary Outcome: Change in LDL-C Concentration From Baseline Over Time Within and Between Treatment Groups
Time Frame: 120 weeks
Population: All subjects were analyzed and contributed LDL-C data for the 'High-Intensity Statin Therapy + RVX000222' and the 'High-Intensity statin therapy + Placebo' arms.
  Subject data is missing across time points.
Measure: Median (Inter-Quartile Range); unit: mmol/L
Arm/Group | High-Intensity Statin Therapy+RVX000222 | High-Intensity Statin Therapy+Placebo
Number analyzed (Participants) | 1212 | 1206
mmol/L
  Baseline: number analyzed (Participants) | 1140 | 1130
  Baseline | 1.690 [1.270 to 2.215] | 1.690 [1.260 to 2.180]
  Visit 11 (Week 24): number analyzed (Participants) | 1005 | 1007
  Visit 11 (Week 24) | 1.530 [1.160 to 2.010] | 1.530 [1.140 to 1.970]
  Visit 14 (Week 52): number analyzed (Participants) | 979 | 986
  Visit 14 (Week 52) | 1.590 [1.210 to 2.120] | 1.655 [1.240 to 2.130]
  Visit 16 Week 76): number analyzed (Participants) | 785 | 799
  Visit 16 Week 76) | 1.600 [1.230 to 2.090] | 1.660 [1.270 to 2.100]
  Visit 18 Week 100): number analyzed (Participants) | 553 | 560
  Visit 18 Week 100) | 1.660 [1.300 to 2.180] | 1.725 [1.300 to 2.220]
  Last Visit on Treatment (LVT): number analyzed (Participants) | 864 | 898
  Last Visit on Treatment (LVT) | 1.700 [1.240 to 2.240] | 1.745 [1.290 to 2.280]
  Follow-up: number analyzed (Participants) | 817 | 839
  Follow-up | 1.650 [1.250 to 2.210] | 1.680 [1.240 to 2.270]

8. Secondary Outcome: Change in HDL-C Concentration From Baseline Over Time Within and Between Treatment Groups
Time Frame: 120 weeks
Population: All subjects were analyzed and contributed HDL-C data for the 'High-Intensity Statin Therapy + RVX000222' and the 'High-Intensity statin therapy + Placebo' arms.
  Subject data is missing across time points.
Measure: Median (Inter-Quartile Range); unit: mmol/L
Arm/Group | High-Intensity Statin Therapy+RVX000222 | High-Intensity Statin Therapy+Placebo
Number analyzed (Participants) | 1212 | 1206
mmol/L
  Baseline: number analyzed (Participants) | 1140 | 1133
  Baseline | 0.870 [0.770 to 0.960] | 0.860 [0.780 to 0.960]
  Visit 11 (Week 24): number analyzed (Participants) | 1005 | 1007
  Visit 11 (Week 24) | 0.970 [0.840 to 1.100] | 0.940 [0.810 to 1.060]
  Visit 14 (Week 52): number analyzed (Participants) | 979 | 986
  Visit 14 (Week 52) | 0.970 [0.840 to 1.110] | 0.930 [0.820 to 1.070]
  Visit 16 Week 76): number analyzed (Participants) | 787 | 800
  Visit 16 Week 76) | 0.960 [0.830 to 1.110] | 0.920 [0.800 to 1.060]
  Visit 18 Week 100) | 0.970 [0.840 to 1.110] | 0.910 [0.810 to 1.060]
  Last Visit on Treatment (LVT): number analyzed (Participants) | 860 | 892
  Last Visit on Treatment (LVT) | 0.990 [0.870 to 1.145] | 0.960 [0.830 to 1.100]
  Follow-up: number analyzed (Participants) | 804 | 823
  Follow-up | 1.010 [0.870 to 1.150] | 0.950 [0.850 to 1.100]

9. Secondary Outcome: Change in Triglyceride (TG) Concentration From Baseline Over Time Within and Between Treatment Groups
Time Frame: 120 weeks
Population: All subjects were analyzed and contributed TG data for the 'High-Intensity Statin Therapy + RVX000222' and the 'High-Intensity statin therapy + Placebo' arms.
  Subject data is missing across time points.
Measure: Median (Inter-Quartile Range); unit: mmol/L
Arm/Group | High-Intensity Statin Therapy+RVX000222 | High-Intensity Statin Therapy+Placebo
Number analyzed (Participants) | 1212 | 1206
mmol/L
  Baseline: number analyzed (Participants) | 1140 | 1132
  Baseline | 1.630 [1.245 to 2.205] | 1.690 [1.310 to 2.275]
  Visit 11 (Week 24): number analyzed (Participants) | 1005 | 1007
  Visit 11 (Week 24) | 1.660 [1.260 to 2.260] | 1.670 [1.200 to 2.270]
  Visit 14 (Week 52): number analyzed (Participants) | 980 | 986
  Visit 14 (Week 52) | 1.735 [1.285 to 2.370] | 1.700 [1.220 to 2.330]
  Visit 16 Week 76): number analyzed (Participants) | 787 | 802
  Visit 16 Week 76) | 1.730 [1.240 to 2.420] | 1.670 [1.200 to 2.330]
  Visit 18 Week 100): number analyzed (Participants) | 554 | 561
  Visit 18 Week 100) | 1.755 [1.260 to 2.420] | 1.610 [1.240 to 2.420]
  Last Visit on Treatment (LVT): number analyzed (Participants) | 865 | 899
  Last Visit on Treatment (LVT) | 1.700 [1.230 to 2.360] | 1.650 [1.210 to 2.330]
  Follow-up: number analyzed (Participants) | 817 | 841
  Follow-up | 1.650 [1.200 to 2.300] | 1.720 [1.270 to 2.380]

10. Secondary Outcome: Change in Hemoglobin (Hb) A1c From Baseline Over Time Within and Between Treatment Groups
Time Frame: 120 weeks
Population: All subjects were analyzed and contributed HbA1c data for the 'High-Intensity Statin Therapy + RVX000222' and the 'High-Intensity statin therapy + Placebo' arms Subject data is missing across time points
Measure: Median (Inter-Quartile Range); unit: % of hemoglobin
Arm/Group | High-Intensity Statin Therapy+RVX000222 | High-Intensity Statin Therapy+Placebo
Number analyzed (Participants) | 1212 | 1207
% of hemoglobin
  Baseline: number analyzed (Participants) | 1202 | 1195
  Baseline | 7.40 [6.40 to 8.70] | 7.30 [6.40 to 8.60]
  Visit 11 (Week 24): number analyzed (Participants) | 1058 | 1048
  Visit 11 (Week 24) | 7.20 [6.40 to 8.50] | 7.20 [6.40 to 8.40]
  Visit 14 (Week 52): number analyzed (Participants) | 1023 | 1037
  Visit 14 (Week 52) | 7.30 [6.40 to 8.60] | 7.30 [6.40 to 8.70]
  Visit 16 (Week 76): number analyzed (Participants) | 808 | 833
  Visit 16 (Week 76) | 7.30 [6.50 to 8.65] | 7.40 [6.50 to 8.60]
  Visit 18 (Week 100): number analyzed (Participants) | 575 | 576
  Visit 18 (Week 100) | 7.30 [6.40 to 8.70] | 7.30 [6.50 to 8.70]
  LVT: number analyzed (Participants) | 900 | 933
  LVT | 7.40 [6.40 to 8.90] | 7.30 [6.40 to 8.70]
  Follow-up: number analyzed (Participants) | 858 | 874
  Follow-up | 7.30 [6.40 to 8.70] | 7.20 [6.40 to 8.60]

11. Secondary Outcome: Change in Glucose From Baseline Over Time Between and Within Treatment Groups
Time Frame: 120 weeks
Population: All subjects were analyzed and contributed glucose data for the 'High-Intensity Statin Therapy + RVX000222' and the 'High-Intensity statin therapy + Placebo' arms.
  Subject data is missing across time points
Measure: Median (Inter-Quartile Range); unit: mmol/L
Arm/Group | High-Intensity Statin Therapy+RVX000222 | High-Intensity Statin Therapy+Placebo
Number analyzed (Participants) | 1212 | 1207
mmol/L
  Baseline: number analyzed (Participants) | 1210 | 1206
  Baseline | 7.590 [6.140 to 9.730] | 7.385 [6.100 to 9.660]
  Visit 11 (Week 24): number analyzed (Participants) | 1068 | 1066
  Visit 11 (Week 24) | 7.925 [6.310 to 10.450] | 7.835 [6.230 to 10.240]
  Visit 14 (Week 52): number analyzed (Participants) | 1030 | 1044
  Visit 14 (Week 52) | 7.900 [6.290 to 10.390] | 7.800 [6.420 to 10.345]
  Visit 16 (Week 76): number analyzed (Participants) | 826 | 844
  Visit 16 (Week 76) | 7.920 [6.390 to 10.340] | 7.840 [6.250 to 10.430]
  Visit 18 (Week 100): number analyzed (Participants) | 580 | 586
  Visit 18 (Week 100) | 8.010 [6.365 to 10.535] | 7.890 [6.280 to 10.670]
  LVT: number analyzed (Participants) | 905 | 940
  LVT | 8.100 [6.440 to 10.750] | 7.795 [6.180 to 10.445]
  Follow-up: number analyzed (Participants) | 860 | 882
  Follow-up | 7.650 [6.250 to 10.130] | 7.595 [6.080 to 10.110]

12. Secondary Outcome: Change in Alkaline Phosphatase (ALP) From Baseline Over Time Within and Between Treatment Groups
Time Frame: 172 weeks
Population: Subject data is missing across time points
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | High-Intensity Statin Therapy+RVX000222 | High-Intensity Statin Therapy+Placebo
Number analyzed (Participants) | 1212 | 1207
U/L
  Baseline | 78.0 [64.0 to 95.5] | 77.0 [64.0 to 93.0]
  Visit 3 (Week 2): number analyzed (Participants) | 1156 | 1151
  Visit 3 (Week 2) | 71.0 [58.0 to 88.0] | 76.0 [62.0 to 91.0]
  Visit 4 (Week 4): number analyzed (Participants) | 1136 | 1131
  Visit 4 (Week 4) | 70.0 [58.0 to 88.0] | 75.0 [63.0 to 92.0]
  Visit 5 (Week 6): number analyzed (Participants) | 1102 | 1108
  Visit 5 (Week 6) | 70.0 [56.0 to 87.0] | 75.0 [61.0 to 93.0]
  Visit 6 (Week 8): number analyzed (Participants) | 1125 | 1098
  Visit 6 (Week 8) | 69.0 [56.0 to 86.0] | 76.0 [62.0 to 92.0]
  Visit 7 (Week 10): number analyzed (Participants) | 1100 | 1095
  Visit 7 (Week 10) | 69.0 [56.0 to 86.0] | 75.0 [62.0 to 92.0]
  Visit 8 (Week 12): number analyzed (Participants) | 1120 | 1109
  Visit 8 (Week 12) | 69.0 [56.0 to 87.0] | 75.0 [62.0 to 93.0]
  Visit 9 (Week 16): number analyzed (Participants) | 1094 | 1095
  Visit 9 (Week 16) | 68.0 [55.0 to 85.0] | 75.0 [61.0 to 92.0]
  Visit 10 (Week 20): number analyzed (Participants) | 1091 | 1081
  Visit 10 (Week 20) | 68.0 [55.0 to 86.0] | 74.0 [61.0 to 92.0]
  Visit 11 (Week 24): number analyzed (Participants) | 1082 | 1070
  Visit 11 (Week 24) | 68.0 [55.0 to 84.0] | 75.0 [60.0 to 92.0]
  Visit 12 (Week 28): number analyzed (Participants) | 1073 | 1079
  Visit 12 (Week 28) | 69.0 [55.0 to 85.0] | 74.0 [61.0 to 93.0]
  Visit 13 (Week 40): number analyzed (Participants) | 1062 | 1068
  Visit 13 (Week 40) | 69.0 [56.0 to 87.0] | 74.0 [61.0 to 93.0]
  Visit 14 (Week 52): number analyzed (Participants) | 1035 | 1047
  Visit 14 (Week 52) | 71.0 [57.0 to 89.0] | 76.0 [61.0 to 96.0]
  Visit 15 (Week 64): number analyzed (Participants) | 965 | 984
  Visit 15 (Week 64) | 71.0 [57.0 to 87.0] | 74.5 [62.0 to 95.5]
  Visit 16 (Week 76): number analyzed (Participants) | 829 | 846
  Visit 16 (Week 76) | 70.0 [58.0 to 88.0] | 76.0 [61.0 to 93.0]
  Visit 17 (Week 88): number analyzed (Participants) | 698 | 717
  Visit 17 (Week 88) | 72.0 [58.0 to 91.0] | 76.0 [62.0 to 95.0]
  Visit 18 (Week 100): number analyzed (Participants) | 580 | 590
  Visit 18 (Week 100) | 72.0 [59.0 to 92.0] | 75.0 [62.0 to 95.0]
  Visit 19 (Week 112): number analyzed (Participants) | 471 | 471
  Visit 19 (Week 112) | 71.0 [58.0 to 90.0] | 75.0 [62.0 to 96.0]
  Visit 20 (Week 124): number analyzed (Participants) | 359 | 357
  Visit 20 (Week 124) | 71.0 [57.0 to 92.0] | 77.0 [63.0 to 95.0]
  Visit 21 (Week 136): number analyzed (Participants) | 228 | 211
  Visit 21 (Week 136) | 69.5 [56.0 to 92.0] | 77.0 [62.0 to 93.0]
  Visit 22 (Week 148): number analyzed (Participants) | 109 | 123
  Visit 22 (Week 148) | 69.0 [56.0 to 88.0] | 76.0 [64.0 to 91.0]
  Visit 23 (Week 160): number analyzed (Participants) | 32 | 30
  Visit 23 (Week 160) | 68.0 [57.5 to 87.5] | 78.0 [55.0 to 89.0]
  Visit 24 (Week 172): number analyzed (Participants) | 2 | 5
  Visit 24 (Week 172) | 75.5 [62.0 to 89.0] | 83.0 [64.0 to 112.0]
  Last Visit on Treatment (LVT): number analyzed (Participants) | 906 | 940
  Last Visit on Treatment (LVT) | 72.0 [59.0 to 91.0] | 77.0 [62.0 to 97.0]
  Follow-up: number analyzed (Participants) | 860 | 882
  Follow-up | 76.0 [63.0 to 93.0] | 76.0 [62.0 to 95.0]

13. Secondary Outcome: Change in C Reactive Protein (CRP) Concentration From Baseline Over Time Within and Between Treatment Groups
Time Frame: 52 weeks
Population: A select subset of subjects in two countries were analyzed for CRP, Subject data is missing across time points.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | High-Intensity Statin Therapy+RVX000222 | High-Intensity Statin Therapy+Placebo
Number analyzed (Participants) | 244 | 239
mg/dL
  Baseline | 2.875 [1.245 to 5.915] | 2.740 [1.130 to 6.150]
  Visit 8 (Week 12): number analyzed (Participants) | 224 | 218
  Visit 8 (Week 12) | 1.755 [0.875 to 3.895] | 1.805 [1.000 to 4.300]
  Visit 14 (Week 52): number analyzed (Participants) | 206 | 201
  Visit 14 (Week 52) | 1.710 [0.860 to 4.050] | 1.580 [0.720 to 3.710]

14. Secondary Outcome: Change in Estimated Glomerular Filtration Rate (eGFR) From Baseline Over Time Within and Between Treatment Groups for Subjects With Impaired Renal Function at Baseline (eGFR <60 mL/Min/1.7m2)
Time Frame: 120 weeks
Population: Subject data is missing across time points
Measure: Median (Inter-Quartile Range); unit: ml/min
Arm/Group | High-Intensity Statin Therapy+RVX000222 | High-Intensity Statin Therapy+Placebo
Number analyzed (Participants) | 121 | 162
ml/min
  Baseline | 51.4 [41.4 to 56.0] | 48.9 [40.6 to 55.9]
  Visit 11 (Week 24): number analyzed (Participants) | 106 | 133
  Visit 11 (Week 24) | 53.0 [41.5 to 63.7] | 53.3 [41.4 to 63.2]
  Visit 14 (Week 52): number analyzed (Participants) | 98 | 126
  Visit 14 (Week 52) | 52.4 [41.3 to 62.2] | 52.5 [41.8 to 63.0]
  Visit 16 (Week 76): number analyzed (Participants) | 80 | 97
  Visit 16 (Week 76) | 50.8 [37.5 to 63.6] | 54.8 [42.5 to 63.8]
  Visit 18 (Week 100): number analyzed (Participants) | 80 | 66
  Visit 18 (Week 100) | 46.5 [34.0 to 59.3] | 56.7 [42.4 to 66.0]
  LVT: number analyzed (Participants) | 87 | 107
  LVT | 52.5 [39.2 to 62.3] | 53.9 [43.3 to 61.1]

15. Post Hoc Outcome: Incidence of First Occurrence of Adjudication-Confirmed Four-Point MACE
Description: First occurrence of four-point MACE defined as a single composite endpoint of cardiovascular (CV) death (including undetermined cause of death) or non-fatal myocardial infarction (MI), stroke or hospital admission for congestive heart failure.
Time Frame: 120 weeks
Measure: Number; unit: events
Arm/Group | High-Intensity Statin Therapy+RVX000222 | High-Intensity Statin Therapy+Placebo
Number analyzed (Participants) | 1212 | 1206
events
  CV Death (CVD) | 45 | 55
  Non-fatal MI | 77 | 94
  Stroke | 17 | 17
  First Hospitalization for CHF | 29 | 48
Statistical Analysis 1: Comparison: High-Intensity Statin Therapy+RVX000222 vs High-Intensity Statin Therapy+Placebo; Test type: Superiority; p = 0.03, Log Rank; Cox Proportional Hazard = 0.78, 95% CI 2-sided [0.63 to 0.98]

ADVERSE EVENTS:
Time Frame: 120 weeks
Arm/Group | High-Intensity Statin Therapy+RVX000222 | High-Intensity Statin Therapy+Placebo
All-Cause Mortality (participants affected / at risk) | 61/1212 | 72/1207
Serious Adverse Events (participants affected / at risk) | 354/1212 | 339/1207
Other Adverse Events (participants affected / at risk) | 830/1212 | 820/1207
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High-Intensity Statin Therapy+RVX000222 (N=1212) | High-Intensity Statin Therapy+Placebo (N=1207)
Angina unstable (Cardiac disorders) | 57 | 39
Acute myocardial infarction (Cardiac disorders) | 42 | 49
Angina pectoris (Cardiac disorders) | 32 | 32
Cardiac failure (Cardiac disorders) | 11 | 28
Myocardial infarction (Cardiac disorders) | 14 | 11
Atrial fibrillation (Cardiac disorders) | 10 | 10
Cardiac failure congestive (Cardiac disorders) | 6 | 9
Coronary artery disease (Cardiac disorders) | 9 | 6
Acute coronary syndrome (Cardiac disorders) | 5 | 9
Cardiac failure acute (Cardiac disorders) | 8 | 6
Coronary artery stenosis (Cardiac disorders) | 5 | 4
Myocardial ischemia (Cardiac disorders) | 5 | 3
Cardiac failure chronic (Cardiac disorders) | 2 | 5
Cardiac arrest (Cardiac disorders) | 1 | 5
Cardiogenic shock (Cardiac disorders) | 2 | 4
Atrial flutter (Cardiac disorders) | 3 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 2 | 2
Ventricular tachycardia (Cardiac disorders) | 3 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 3
Supraventricular tachycardia (Cardiac disorders) | 0 | 3
Ventricular fibrillation (Cardiac disorders) | 1 | 2
Coronary artery occlusion (Cardiac disorders) | 0 | 2
Left ventricular failure (Cardiac disorders) | 2 | 0
Mitral valve incompetence (Cardiac disorders) | 2 | 0
Anginal equivalent (Cardiac disorders) | 0 | 1
Aortic valve incompetence (Cardiac disorders) | 1 | 0
Aortic valve stenosis (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 1
Atrioventricular block (Cardiac disorders) | 1 | 0
Bradyarrhythmia (Cardiac disorders) | 0 | 1
Cardiac discomfort (Cardiac disorders) | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Intracardiac thrombus (Cardiac disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 1
Microvascular coronary artery disease (Cardiac disorders) | 1 | 0
Myocardial fibrosis (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 1
Sinus node dysfunction (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Ventricular arrhythmia (Cardiac disorders) | 0 | 1
Ventricular failure (Cardiac disorders) | 0 | 1
Pneumonia (Infections and infestations) | 15 | 17
Urinary tract infection (Infections and infestations) | 6 | 3
Cellulitis (Infections and infestations) | 2 | 3
Bronchitis (Infections and infestations) | 2 | 4
Osteomyelitis (Infections and infestations) | 3 | 2
Gangrene (Infections and infestations) | 3 | 1
Sepsis (Infections and infestations) | 2 | 2
Septic shock (Infections and infestations) | 3 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 2
Viral infection (Infections and infestations) | 3 | 1
Diverticulitis (Infections and infestations) | 1 | 2
Ertsipelas (Infections and infestations) | 2 | 1
Gastroenteritis (Infections and infestations) | 2 | 1
Urosepsis (Infections and infestations) | 2 | 1
Diabetic gangrene (Infections and infestations) | 1 | 1
Escherichia urinary tract infection (Infections and infestations) | 2 | 0
Postoperative wound infection (Infections and infestations) | 2 | 0
Pyelonephritis (Infections and infestations) | 1 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 2
Acute endocarditis (Infections and infestations) | 1 | 0
Anal abscess (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Appendicitis perforated (Infections and infestations) | 1 | 0
Brain abscess (Infections and infestations) | 1 | 0
Cholecystitis infective (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 0
Diabetic foot infection (Infections and infestations) | 0 | 1
Gallbladder empyema (Infections and infestations) | 1 | 0
Hepatitis E (Infections and infestations) | 1 | 0
Hepatitis viral (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 0 | 1
Mastoiditis (Infections and infestations) | 0 | 1
Mediastinitis (Infections and infestations) | 1 | 0
Necrotising fasciitis (Infections and infestations) | 0 | 1
Opportunistic infection (Infections and infestations) | 0 | 1
Pneumonia legionella (Infections and infestations) | 0 | 1
Pneumonia necrotising (Infections and infestations) | 1 | 0
Pneumonia streptococcal (Infections and infestations) | 0 | 1
Scrotal abscess (Infections and infestations) | 1 | 0
Soft tissue infection (Infections and infestations) | 0 | 1
Staphylococcal skin infection (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 1
Urinary tract infection bacterial (Infections and infestations) | 0 | 1
Urinary tract infection enterococcal (Infections and infestations) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 5 | 5
Cerebrovascular accident (Nervous system disorders) | 4 | 2
Syncope (Infections and infestations) | 1 | 5
Transient ischaemic attack (Infections and infestations) | 3 | 3
Carotid artery stenosis (Nervous system disorders) | 2 | 2
Cerebral infarction (Nervous system disorders) | 2 | 2
Haemorrhagic stroke (Nervous system disorders) | 1 | 1
Quadriparesis (Nervous system disorders) | 2 | 0
VIIth nerve paralysis (Nervous system disorders) | 1 | 1
Brain stem stroke (Nervous system disorders) | 0 | 1
Carotid sinus syndrome (Nervous system disorders) | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1
Cerebral arteriosclerosis (Nervous system disorders) | 0 | 1
Cervical cord compression (Nervous system disorders) | 1 | 0
Diabetic neuropathy (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Dysarthria (Nervous system disorders) | 1 | 0
Febrile convulsion (Nervous system disorders) | 1 | 0
Guillain-Barre syndrome (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Intracranial aneurysm (Nervous system disorders) | 1 | 0
Lumbar radiculopathy (Nervous system disorders) | 1 | 0
Lumbosacral radiculopathy (Nervous system disorders) | 1 | 0
Nerve compression (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1
Parkinson's disease (Nervous system disorders) | 1 | 0
Polyneuropathy (Nervous system disorders) | 0 | 1
Psychomotor hyperactivity (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 33 | 25
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 2
Gastritis erosive (Gastrointestinal disorders) | 2 | 2
Inguinal hernia (Gastrointestinal disorders) | 3 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 2
Anal fissure (Gastrointestinal disorders) | 2 | 0
Chronic gastritis (Gastrointestinal disorders) | 1 | 1
Gastric polyps (Gastrointestinal disorders) | 1 | 1
Gastritis (Gastrointestinal disorders) | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 1
Large intestine polyp (Gastrointestinal disorders) | 1 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Acute abdomen (Gastrointestinal disorders) | 0 | 1
Diabetic gastroparesis (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 0 | 1
Gastrointestinal angiodysplasia haemorrhagic (Gastrointestinal disorders) | 0 | 1
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 0 | 1
Haemorrhoids thrombosed (Gastrointestinal disorders) | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Oesophageal obstruction (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 | 0
Salivary gland calculus (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 7 | 7
Hypertension (Vascular disorders) | 2 | 9
Hypertensive crisis (Vascular disorders) | 1 | 7
Hypertensive emergency (Vascular disorders) | 2 | 2
Aortic stenosis (Vascular disorders) | 1 | 2
Peripheral ischaemia (Vascular disorders) | 2 | 1
Hypotension (Vascular disorders) | 2 | 0
Hypovolaemic shock (Vascular disorders) | 1 | 1
Arteriosclerosis (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Extremity necrosis (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 0 | 1
Ischaemia (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0
Peripheral artery stenosis (Vascular disorders) | 1 | 0
Peripheral artery thrombosis (Vascular disorders) | 1 | 0
Subclavian artery occlusion (Vascular disorders) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Benign hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung squamous cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Nasopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oropharyngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Small cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-cardiac chest pain (General disorders) | 10 | 12
Sudden death (General disorders) | 2 | 6
Death (General disorders) | 3 | 3
Sudden cardiac death (General disorders) | 0 | 3
Pyrexia (General disorders) | 2 | 0
Vascular stent restenosis (General disorders) | 0 | 2
Chest pain (General disorders) | 1 | 0
Exercise tolerance decreased (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Vascular stent occlusion (General disorders) | 0 | 1
Vascular stent stenosis (General disorders) | 1 | 0
Vascular stent thrombosis (General disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 9 | 7
Chronic kidney disease (Renal and urinary disorders) | 4 | 3
Nephrolithiasis (Renal and urinary disorders) | 2 | 2
Renal failure (Renal and urinary disorders) | 2 | 2
Calculus ureteric (Renal and urinary disorders) | 2 | 1
Ureteric stenosis (Renal and urinary disorders) | 1 | 2
Diabetic nephropathy (Renal and urinary disorders) | 0 | 2
Urinary retention (Renal and urinary disorders) | 0 | 2
Azotaemia (Renal and urinary disorders) | 0 | 1
Bladder perforation (Renal and urinary disorders) | 1 | 0
Calculus bladder (Renal and urinary disorders) | 1 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Nephropathy (Renal and urinary disorders) | 1 | 0
Renal artery stenosis (Renal and urinary disorders) | 0 | 1
Renal mass (Renal and urinary disorders) | 1 | 0
Ureteric rupture (Renal and urinary disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 7 | 9
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Paranasal sinus haematoma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus polyp (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Vocal cord cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 1
Coronary artery restenosis (Injury, poisoning and procedural complications) | 1 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 1
Hip fracture (Injury, poisoning and procedural complications) | 2 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 2
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 1
Brain contusion (Injury, poisoning and procedural complications) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Lumbosacral plexus injury (Injury, poisoning and procedural complications) | 0 | 1
Nerve root injury (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Postpericardiotomy syndrome (Injury, poisoning and procedural complications) | 1 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 1
Radial head dislocation (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Skull fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 6 | 5
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 2
Metabolic disorder (Metabolism and nutrition disorders) | 1 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 5
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1
Hepatic lesion (Hepatobiliary disorders) | 1 | 0
Hepatitis acute (Hepatobiliary disorders) | 0 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 1
Cataract (Eye disorders) | 2 | 2
Glaucoma (Eye disorders) | 0 | 3
Diabetic retinopathy (Eye disorders) | 1 | 1
Detachment of retinal pigment epithelium (Eye disorders) | 0 | 1
Eye haemorrhage (Eye disorders) | 1 | 0
Hypotony of eye (Eye disorders) | 0 | 1
Iris bombe (Eye disorders) | 0 | 1
Posterior capsule opacification (Eye disorders) | 0 | 1
Retinal detachment (Eye disorders) | 0 | 1
Vitreous haemorrhage (Eye disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 4 | 1
Hypochromic anaemia (Blood and lymphatic system disorders) | 2 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1
Hepatic enzyme increased (Investigations) | 3 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Blood pressure abnormal (Investigations) | 1 | 0
Depression (Psychiatric disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Anxiety disorder (Psychiatric disorders) | 1 | 0
Completed suicide (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 2 | 2
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 1 | 0
Amyloidosis (Immune system disorders) | 0 | 1
Medical device removal (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | High-Intensity Statin Therapy+RVX000222 (N=1212) | High-Intensity Statin Therapy+Placebo (N=1207)
Nasopharyngitis (Infections and infestations) | 46 | 56
Urinary tract infection (Infections and infestations) | 58 | 40
Influenza (Infections and infestations) | 43 | 47
Bronchitis (Infections and infestations) | 25 | 32
Pneumonia (Infections and infestations) | 27 | 26
Upper respiratory tract infection (Infections and infestations) | 29 | 24
Angina (Cardiac disorders) | 74 | 76
Angina unstable (Cardiac disorders) | 58 | 41
Acute myocardial infarction (Cardiac disorders) | 42 | 50
Cardiac failure (Cardiac disorders) | 22 | 38
Diarrhoea (Gastrointestinal disorders) | 43 | 44
Abdominal pain (Gastrointestinal disorders) | 12 | 24
Nausea (Gastrointestinal disorders) | 26 | 7
Hepatobiliary (Gastrointestinal disorders) | 24 | 42
Myalgia (Musculoskeletal and connective tissue disorders) | 37 | 33
Back pain (Musculoskeletal and connective tissue disorders) | 27 | 28
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15 | 26
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 24
Worsening diabetes mellitus (Metabolism and nutrition disorders) | 93 | 93
Hypertension (Vascular disorders) | 72 | 72
ALT increase (Investigations) | 64 | 18
Non-cardiac chest pain (General disorders) | 33 | 39
Anemia (Blood and lymphatic system disorders) | 36 | 40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-10-31): https://cdn.clinicaltrials.gov/large-docs/55/NCT02586155/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-10): https://cdn.clinicaltrials.gov/large-docs/55/NCT02586155/SAP_001.pdf